CLINICAL TRIAL: NCT02500914
Title: A Phase 1a/1b Dose Escalation and Expansion Study of Single-agent SC-002 in Subjects With Relapsed or Refractory Small Cell Lung Cancer and Large Cell Neuroendocrine Carcinoma
Brief Title: SC-002 in Small Cell Lung Cancer and Large Cell Neuroendocrine Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Considerations
Sponsor: Stemcentrx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRX002-001
Record Dates: First submitted 2015-07-06; First posted 2015-07-17 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Small Cell Lung Cancer
Keywords: small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — SC002

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SC-002 (Experimental): Part 1A (Dose Escalation) - IV infusion; safety data will be reviewed prior to dose escalation decision. Dose escalation will complete when recommended dose (RD) is determined. RD will be the maximum tolerated dose (MTD) or lower dose that provides adequate PK exposure, immunogenicity, and preliminary evidence of antitumor activity with tolerability.
  Part 1B (Dose Expansion) - IV infusion; once MTD and/or RD has been determined in Part 1A, an expansion cohort of approximately 60 patients with SCLC or LCNEC will be enrolled to further characterize the safety profile and clinical activity of the RD. Patients may continue treatment until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: SC-002

INTERVENTIONS:
Drug: SC-002 — SC-002 will be administered by IV infusion over approximately 30 minutes every 3 weeks

SUMMARY:
This is a Phase 1a/1b study of SC-002 in patients with relapsed small cell lung cancer (SCLC) or large cell neuroendocrine carcinoma (LCNEC). SC-002 is an antibody-drug conjugate (ADC) comprised of a monoclonal antibody linked to a potent chemotherapy.

The purpose of this study is to assess the safety and tolerability of SC-002 at different dose levels, to determine the highest dose of SC-002 that can be given to patients with SCLC or LCNEC, to evaluate the side effects of SC-002, and to assess the anti-cancer activity of SC-002.

DETAILED DESCRIPTION:
Part 1A is a dose escalation study in patients with small cell lung cancer or large cell neuroendocrine carcinoma with cytologically confirmed, limited or extensive SCLC or LCNEC that have relapsed or refractory limited or extensive disease following no more than 2 prior chemotherapy regimens.

Part 1B is an expansion study where patients will be enrolled and treated in order to further characterize safety and preliminary efficacy in patients with SCLC or LCNEC and further characterize PK, immunogenicity and target expression and possible relationship to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC (either limited or extensive disease) or LCNEC, that has relapsed from the most current treatment or was refractory to treatment
* Evidence of progressive disease during or following no more than 2 prior chemotherapy regimens
* Measurable disease as defined by RECIST
* ECOG performance status of 0 or 1
* Adequate hematological and organ function as confirmed by laboratory values
* Treatment with anticancer/investigational drugs, therapy ≤ 4 weeks prior to first dose of SC-002

Exclusion Criteria:

* Active central nervous system metastases
* Uncontrolled cardiac disease
* Positive serology for hepatitis B or hepatitis C or known HIV infection
* Presence of any condition that may increase the risks associated with study participation and interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-06; Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
Number of subjects with adverse events as a measure of safety and tolerability | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics of SC-002 | Cycle 1 and 4: days 1, 2, 4, 8, 15; Cycles 2, 3, and 5: day 1 only
  Standard PK variables to be assessed include AUC, Tmax, Cmax, Ctrough, T1/2, CL, Vss
RECIST v1.1 assessed objective response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lawrence, D.O., Study Director — Novella Clinical
Locations (4):
- United States (4):
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - New York, New York
  - Nashville, Tennessee

REFERENCES:
- [Derived] Morgensztern D, Johnson M, Rudin CM, Rossi M, Lazarov M, Brickman D, Fong A. SC-002 in patients with relapsed or refractory small cell lung cancer and large cell neuroendocrine carcinoma: Phase 1 study. Lung Cancer. 2020 Jul;145:126-131. doi: 10.1016/j.lungcan.2020.04.017. Epub 2020 May 12. PMID 32438272